CLINICAL TRIAL: NCT00954538
Title: A Three Part Study to Evaluate the Safety, Radiation Dosimetry, Biokinetics, and Effectiveness of [18F]MK-3328, a Radiotracer for Use in Positron Emission Tomography
Brief Title: Safety, Radiation Dosimetry, Biokinetics, and Effectiveness of [18F]MK3328 (MK-3328-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 3328-001; 2009_630 (Other: Merck Registration Number)
Record Dates: First submitted 2009-08-06; First posted 2009-08-07 (Estimated); Results first posted 2014-02-05 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part I, Healthy Participants (Experimental): Healthy participants will receive a single intravenous (IV) dose of ~150 megabecquerel (MBq) [18F]MK-3328 in Part I of the study
  Interventions: Drug: [18F]MK-3328
- Part II, HE and AD Participants (Experimental): HE and AD participants will receive a single IV dose of ~150 megabecquerel (MBq) [18F]MK-3328 in Part II of the study
  Interventions: Drug: [18F]MK-3328
- Part III, HE and AD Participants (Experimental): HE and AD participants will receive two separate IV doses of ~150 megabecquerel (MBq) [18F]MK-3328 in Part III of the study
  Interventions: Drug: [18F]MK-3328

INTERVENTIONS:
Drug: [18F]MK-3328 — IV dose of ~150 megabecquerel (MBq) [18F]MK-3328

SUMMARY:
This study will estimate the radiochemical and radiation safety and assess the efficacy of [18F]MK-3328, a novel positron emission tomography (PET) tracer. The study safety hypotheses will test whether [18F]MK-3328 is sufficiently safe and well-tolerated, based on an assessment of clinical and laboratory evaluations and adverse experiences in healthy participants, including healthy elderly (HE) participants, and Alzheimer's disease (AD) participants, to permit continued investigation. The study efficacy hypothesis will test whether [18F]MK-3328 can discriminate between AD participants and cognitively normal elderly control participants based on tracer volume of distribution, or one of its surrogates, in brain posterior cingulate gyrus.

ELIGIBILITY:
Inclusion Criteria:

Part I:

* Participant is male or female of non-reproductive potential between 50 and 65 years old.
* Participant is less than 6'5" tall
* Participant is in good health
* Participant has been a non-smoker for at least 10 years

Parts II and III:

* Male or female of non-reproductive potential at least 55 years of age
* Participant is cognitively normal (HE participants), or has probable mild-to moderate AD (AD participants)
* Participant is willing to have an arterial catheter placed in the radial artery (Part II only)

Exclusion Criteria:

Part I:

* Participant has a history of stroke, seizures, or neurological disorder
* Participant has or has a history of any disease or condition, or takes any medication that would interfere with assessment of the tracer or make participation unsafe or unduly uncomfortable

Parts II and III:

* Participant has a history or current evidence of any neurological or neurodegenerative disorder other than AD that is associated with altered cognition
* Participant has or has a history of any disease or condition, or takes any medication that would interfere with assessment of the tracer or make participation unsafe or unduly uncomfortable
* Participant is living in a nursing home or skilled nursing facility

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2009-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Participants (Part I Only): Healthy participants received a single intravenous (IV) dose of ~150 megabecquerel (MBq) [18F]MK-3328, followed by Positron Emission Tomography (PET) imaging of the whole body (Part I)
- Healthy Elderly (HE) Participants (Part II Only): HE participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain (Part II)
- Alzheimer's Disease (AD) Participants (Part II Only): AD participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain (Part II)
- HE Participants (Part III Only): HE participants received up to two separate IV doses of ~150 MBq [18F]MK-3328; each dose was followed by PET imaging of the brain (Part III)
- AD Participants (Part III Only): AD participants received up to two separate IV doses of ~150 MBq [18F]MK-3328; each dose was followed by PET imaging of the brain (Part III)
- HE Participants (Part II + III): HE participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain (Part II) / HE Participants who completed Part II could receive a second IV dose of ~150 MBq [18F]MK-3328 in Part III; this dose was followed by PET imaging of the brain
Period: Part I
Arm/Group | Healthy Participants (Part I Only) | Healthy Elderly (HE) Participants (Part II Only) | Alzheimer's Disease (AD) Participants (Part II Only) | HE Participants (Part III Only) | AD Participants (Part III Only) | HE Participants (Part II + III)
Started | 3 (These subjects did not participate in Part II or III) | 0 | 0 | 0 | 0 | 0
Completed | 3 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part II
Arm/Group | Healthy Participants (Part I Only) | Healthy Elderly (HE) Participants (Part II Only) | Alzheimer's Disease (AD) Participants (Part II Only) | HE Participants (Part III Only) | AD Participants (Part III Only) | HE Participants (Part II + III)
Started | 0 | 1 (This subject did not participate in Part I or III) | 3 (These subjects did not participate in Part I or III) | 0 | 0 | 2 (These subjects did not participate in Part I and did participate in Part II and III)
Completed | 0 | 1 | 3 | 0 | 0 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Part III
Arm/Group | Healthy Participants (Part I Only) | Healthy Elderly (HE) Participants (Part II Only) | Alzheimer's Disease (AD) Participants (Part II Only) | HE Participants (Part III Only) | AD Participants (Part III Only) | HE Participants (Part II + III)
Started | 0 | 0 | 0 | 4 (These subjects did not participate in Part I or II) | 6 (These subjects did not participate in Part I or II) | 2 (These subjects did not participate in Part I and did participate in Part II and III)
Completed | 0 | 0 | 0 | 4 | 5 (The subject who did not complete received 1 dose of study drug) | 2
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Healthy Participants (Part I) + HE Participants (Part II/III): This group includes Healthy participants (Part I) and HE participants (Part II/III). Participants were administered one or two IV doses of ~150 MBq [18F]MK-3328; all doses were followed by PET imaging of whole body or brain
- AD Participants (Part II/III): This group includes AD participants (Part II/III). Participants were administered one or two IV doses of ~150 MBq [18F]MK-3328; all doses were followed by PET imaging of brain
- Total: Total of all reporting groups
Arm/Group | Healthy Participants (Part I) + HE Participants (Part II/III) | AD Participants (Part II/III) | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (6.3) | 70.7 (5.5) | 65.8 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Adverse Event (AE)
Description: An AE is any unfavorable and unintended change in the structure, function or chemistry of the body temporally associated with study drug administration, whether or not considered related to the study drug.
Time Frame: Up to 14 days after last dose
Population: All participants who received [18F]MK-3328
Measure: Number; unit: participants
Groups:
- All Study Participants: Participants were administered one or two IV doses of ~150 MBq [18F]MK-3328; all doses were followed by PET imaging of whole body or brain
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
participants | 8

2. Primary Outcome: Number of Participants Who Discontinued Study Due to an AE
Description: as for outcome 1
Time Frame: Up to 14 days after last dose
Population: All participants who received [18F]MK-3328
Measure: Number; unit: participants
Arm/Group | All Study Participants
Number analyzed (Participants) | 19
participants | 0

3. Primary Outcome: Effective Dose of [18F]MK-3328
Description: Using PET whole body images acquired after dosing, regions of interest (ROIs) were drawn in all organs showing visible [18F]MK-3328 accumulation. Time activity curves (TACs) showing total [18F]MK-3328 retention as a function of time were determined for each organ. Residence times were calculated from the area under each organ TAC. Radiation exposure of the body and critical organs was calculated from the [18F]MK-3328 residence times using OLINDA (Organ Level Internal Dose Assessment) software. For each organ, the equivalent dose, which is the absorbed radiation dose weighted for the degree of the biological effect of different types of radiation, was calculated. The total radiation exposure to the body is expressed as the effective dose, which is the sum of the equivalent doses in each organ multiplied by a weighting factor for the type of tissue exposed. Effective dose is the primary surrogate for radiation risk. The unit of effective dose is the Sievert (Sv).
Time Frame: Up to approximately 6 hours post dose
Population: All participants who received [18F]MK-3328 in Part I of study
Measure: Mean (Standard Deviation); unit: µSv/MBq
Groups:
- Healthy Participants (Part I): Healthy participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the whole body (Part I)
Arm/Group | Healthy Participants (Part I)
Number analyzed (Participants) | 3
µSv/MBq | 18.2 (2.0)

4. Primary Outcome: Organ Effective Dose of [18F]MK-3328
Description: Using PET whole body images acquired after dosing, ROIs were drawn in all organs showing visible [18F]MK-3328 accumulation. TACs showing total [18F]MK-3328 retention as a function of time were determined for each organ. Residence times were calculated from the area under each organ TAC. Radiation exposure of the body and critical organs was calculated from the [18F]MK-3328 residence times using OLINDA software. For each organ, the equivalent dose, which is the absorbed radiation dose weighted for the degree of the biological effect of different types of radiation, was calculated. The organ effective dose is the equivalent dose in each organ multiplied by a weighting factor for the type of tissue exposed. The unit of organ effective dose is Sv.
Time Frame: Up to approximately 6 hours post dose
Population: All participants who received [18F]MK-3328 in Part I of study
Measure: Mean (Standard Deviation); unit: µSv/MBq
Arm/Group | Healthy Participants (Part I)
Number analyzed (Participants) | 3
µSv/MBq
  Adrenals | 0.0404 (0.0147)
  Brain | 0.0635 (0.0192)
  Breasts | 0.307 (0.0468)
  Gallbladder Wall | 0 (0)
  Lower Large Intestine Wall | 2.57 (0.101)
  Small Intestine | 0.149 (0.0716)
  Stomach Wall | 1.25 (0.195)
  Upper Large Intestine Wall | 0.519 (0.577)
  Heart Wall | 0 (0)
  Kidneys | 0.963 (1.38)
  Liver | 1.35 (0.302)
  Lungs | 1.71 (0.204)
  Muscle | 0.0268 (0.0103)
  Ovaries | 3.06 (0.226)
  Pancreas | 0.0399 (0.0152)
  Red Marrow | 2.36 (0.265)
  Osteogenic Cells | 0.181 (0.0200)
  Skin | 0.0575 (0.00864)
  Spleen | 0.0445 (0.0133)
  Testes | 0 (0)
  Thymus | 0.0247 (0.00904)
  Thyroid | 0.675 (0.0864)
  Urinary Bladder Wall | 2.75 (0.598)
  Uterus | 0.0502 (0.0229)
  Rest of Body | 0 (0)

5. Primary Outcome: Mean Brain Cortical [18F]MK-3328 Standard Uptake Value Ratio (SUVR) in AD Participants and HE Participants
Description: Using PET brain images acquired after dosing, regions of interest (ROIs) were drawn in identified brain areas. The ROIs were projected onto all frames of the dynamic PET scans in order to generate [18F]MK-3328 tissue TACs. SUVR is calculated as the ratio of the average [18F]MK-3328 uptake over 60-90 minutes post dose in the target brain region and the cerebellum. Cortical SUVR is reported, which is a mean SUVR derived from SUVR from multiple brain regions (frontal cortex, parietal cortex, anterior cingulate gyrus, posterior cingulate gyrus, temporal cortex, lateral temporal cortex and occipital cortices).
Time Frame: 60-90 minutes post dose
Population: All participants who received [18F]MK-3328 in Part II of study
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- AD Participants (Part II): AD participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain (Part II)
- HE Participants (Part II): HE participants received a single IV dose of ~150 MBq [18F]MK-3328, followed by PET imaging of the brain (Part II)
Arm/Group | AD Participants (Part II) | HE Participants (Part II)
Number analyzed (Participants) | 3 | 3
ratio | 1.75 (0.14) [1.33 to 1.61] | 1.34 (0.07) [1.23 to 1.48]
Statistical Analysis 1: Comparison: AD Participants (Part II) vs HE Participants (Part II); Test type: Superiority or Other; p < 0.01, t-test, 2 sided

6. Primary Outcome: Least Squares (LS) Mean [18F]MK-3328 SUVR in Brain Posterior Cingulate Gyrus in AD Participants and HE Participants
Description: Using PET brain images acquired after the second dose of [18F]MK-3328, regions of interest (ROIs) were drawn in identified brain areas. The ROIs were projected onto all frames of the dynamic PET scans in order to generate [18F]MK-3328 tissue TACs. Posterior cingulate gyrus SUVR was calculated as the ratio of the average [18F]MK-3328 uptake over 60-90 minutes post dose in the target brain region and the cerebellum.
Time Frame: 60-90 minutes after second dose
Population: All participants who received a second dose of [18F]MK-3328 in Part III of study
Measure: Least Squares Mean (95% Confidence Interval); unit: ratio
Groups:
- AD Participants (Part III): AD participants received two separate IV doses of ~150 MBq [18F]MK-3328; each dose was followed by PET imaging of the brain (Part III)
- HE Participants (Part III): HE participants received two separate IV doses of ~150 MBq [18F]MK-3328; each dose was followed by PET imaging of the brain (Part III)
Arm/Group | AD Participants (Part III) | HE Participants (Part III)
Number analyzed (Participants) | 5 | 6
ratio | 1.47 [1.33 to 1.61] | 1.35 [1.23 to 1.48]
Statistical Analysis 1: Comparison: AD Participants (Part III) vs HE Participants (Part III); A 90% confidence interval was calculated for the group difference (AD - HE) using the model results. As prespecified by the analysis plan, if the lower bound of the 90% confidence interval is above 0, then the hypothesis that [18F]MK-3328 can discriminate between AD patients and cognitively normal elderly controls as measured by regional tracer uptake following single IV doses of [18F]MK-3328 is supported; Test type: Superiority or Other; Linear Fixed Effects Model; LS Mean Difference = 0.12, 90% CI 2-sided [-0.04 to 0.27] — Difference = AD group value - HE group value

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose
Arm/Group | All Study Participants
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 8/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Study Participants (N=19)
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Feeling hot (General disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Dysgeusia (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Sensory loss (Nervous system disorders) | 1
Injection site pain (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission. Sponsor review can be expedited to meet publication guidelines.